CLINICAL TRIAL: NCT06573723
Title: Institutional Registries of Rare Diseases at Hospital Italiano de Buenos Aires (HIBA)
Brief Title: Institutional Registry of Rare Diseases
Status: Recruiting | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, MARIA LOURDES POSADAS MARTINEZ, Principal Investigator, Hospital Italiano de Buenos Aires
Other Study IDs: 7014; 12332 (Registry Identifier: PRIISA)
Record Dates: First submitted 2024-08-06; First posted 2024-08-27 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Rare Diseases; Amyloidosis; Sarcoidosis; Phacomatosis; Pheochromocytoma; Paraganglioma; Von Hippel-Lindau Disease; Immunoglobulin G4-Related Disease; Demyelinating Diseases; Inborn Errors of Metabolism; Eosinophilic Gastrointestinal Disorders; Hypertrophic Cardiomyopathy; Gaucher Disease; Congenital Adrenal Hyperplasia; Hereditary Angioedema; Pulmonary Hypertension; Wilson Disease; Vascular Anomalies; Mastocytosis; Multiple Endocrine Neoplasia; Inflammatory Bowel Diseases; Prader-Willi Syndrome; Hirschsprung Disease; Cushing Syndrome; HHT; Hemorrhagic Hereditary Telangiectasia
Keywords: rare diseases; amyloidosis; sarcoidosis; Phacomatosis; pheochromocytoma; paraganglioma; Von Hippel-Lindau Disease; Immunoglobulin G4-Related Disease; Demyelinating Diseases; Inborn Errors of Metabolism; Eosinophilic Gastrointestinal Disorders; Hypertrophic Cardiomyopathy; Gaucher Disease; Congenital Adrenal Hyperplasia; Hereditary Angioedema; Pulmonary Hypertension; Wilson Disease; Vascular Anomalies; Mastocytosis; Multiple Endocrine Neoplasia; Inflammatory Bowel Diseases; Prader-Willi Syndrome; Hirschsprung Disease; Cushing Syndrome; Hemorrhagic Hereditary Telangiectasia
MeSH Terms: conditions — Rare Diseases; Amyloidosis; Sarcoidosis; Neurocutaneous Syndromes; Pheochromocytoma; Paraganglioma; von Hippel-Lindau Disease; Immunoglobulin G4-Related Disease; Demyelinating Diseases; Metabolism, Inborn Errors; Eosinophilic Esophagitis; Cardiomyopathy, Hypertrophic; Gaucher Disease; Adrenal Hyperplasia, Congenital; Angioedemas, Hereditary; Hypertension, Pulmonary; Hepatolenticular Degeneration; Vascular Malformations; Mastocytosis; Multiple Endocrine Neoplasia; Inflammatory Bowel Diseases; Prader-Willi Syndrome; Hirschsprung Disease; Cushing Syndrome; Telangiectasia, Hereditary Hemorrhagic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — blood and tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to create a single macro registry system with data collection on common clinical features, grouping the different rare diseases (RD).

Moreover, the specific goals are to generate an alert system for possible cases of RD with data from the electronic medical record, to describe the occurrence of RD in the evaluated population, to characterize the population, to describe patterns of diagnosis and treatment of RD present at the time, and to explore patient-reported outcomes.

DETAILED DESCRIPTION:
Rare Diseases (RD) pose a health challenge due to their complexity and low prevalence, generating a burden in terms of morbidity and mortality and costs.

The fragmentation of data on these diseases makes it difficult to understand them comprehensively. Therefore, the creation of a macro institutional registry that brings together information on RD would facilitate research in this field.

The registries are organized systems of systematic data collection of a large number of patients quickly and efficiently on a particular disease at a given time.

The main difficulty of the registries is the guarantee of the quality of their data.

The main objectives of the registry are:

Understand risk factors and prognosis. Evaluate the diagnostic and therapeutic comparison with current standards. Advance knowledge of the disease to optimize the assessment, treatment and monitoring of patients.

Analyze the effectiveness of new therapies. Studying differences between populations. Quickly estimate the morbidity, mortality and resource utilization associated with a disease entity.

Examine the course of a disease Formulate novel hypotheses for further prospective studies.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and/or molecular diagnosis of any of the following rare diseases: Amyloidosis, Sarcoidosis, Phacomatosis, Pheochromocytoma, Paraganglioma, Von Hippel-Lindau Disease, Immunoglobulin G4-Related Disease, Demyelinating Diseases, Inborn Errors of Metabolism, Eosinophilic Gastrointestinal Disorders, Hypertrophic Cardiomyopathy, Gaucher Disease, Congenital Adrenal Hyperplasia, Hereditary Angioedema, Pulmonary Hypertension, Wilson Disease, Vascular Anomalies, Mastocytosis, Multiple Endocrine Neoplasia, Inflammatory Bowel Diseases, Prader-Willi Syndrome, Hirschsprung Disease, or Cushing Syndrome.
* Must be followed at Hospital Italiano de Buenos Aires.

Exclusion Criteria:

- Refusal to participate in the study or in the informed consent process.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People of any age, with a confirmed diagnosis of one or more rare diseases and followed up at Hospital Italiano de Buenos Aires, categorized as such according to the Orpha code from the List of Rare Diseases of the Ministry of Health of the Nation.
Sampling Method: Non-Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2034-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival Rate | From date of enrollment/ diagnosis until the date of death/ last follow up, assessed up to 5 years.
  The overall survival rate will be assessed by calculating the time from the date of enrollment/diagnosis until the date of death from any cause or date of last follow up.
Mortality Rate | From date of enrollment/ diagnosis until the date of death, assessed up to 5 years.
  The mortality rate will be determined by the number of participants who die from any cause during the study period. The data will be reported as the percentage of participants who die within the specified time frame.
Time to First Treatment | From date of diagnosis until the initiation of first treatment, assessed up to 12 months.
  The time to first treatment will be measured from the date of diagnosis until the initiation of the first therapeutic intervention. The data will be summarized as the median time in weeks.
Demographic and Epidemiologic Profile | At baseline, assessed at the time of enrollment.
  Demographic and epidemiologic characteristics, including age, gender, ethnicity, and geographic location, will be described for all participants. The data will be summarized using descriptive statistics.
Clinical Characteristics and Disease Progression | From date of enrollment until the end of the study, assessed up to 5 years.
  Clinical characteristics, including disease stage, comorbidities, and symptoms, will be documented for each participant. Disease progression will be monitored and reported using standardized criteria for each illness.
Treatment Modalities Received | From the initiation of first treatment until the last recorded intervention, assessed up to 5 years.
  Types of treatments received, including medication, surgery, and other therapeutic interventions, will be recorded for each participant. Data will be categorized by treatment type.
Treatment Response | From the initiation of treatment until documented disease progression or treatment cessation, assessed up to 5 years.
  Response to treatment will be evaluated using standardized response criteria for each illness. The data will be reported as the percentage of participants achieving partial or complete response.
Incidence of Treatment-Related Adverse Events | From the initiation of treatment until 12 months after the last dose, assessed up to 5 years.
  The incidence of treatment-related adverse events will be recorded and graded according to CTCAE version 5.0. The data will be reported as the number of participants experiencing adverse events by grade.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Serra, PhD, Principal Investigator — HIBA; Soledad Kleppe, MD, Principal Investigator — HIBA; Maria Lourdes Posadas Martinez, PhD, Principal Investigator — HIBA; Luis Mazzuoccolo, MD, Study Chair — HIBA - dermatología; María Fabiana Russo Picasso, MD, Study Chair — HIBA - endocrinología; Eduardo Jorge Premoli, MD, Study Chair — HIBA - oftalmología; Mariano Martín Marcolongo, MD, Study Chair — HIBA - gastroenterología; Javier Pollan, MD, Study Chair — HIBA - clínica médica; Adrian Gadano, MD, Study Chair — HIBA - investigación; Pablo Lobos, MD, Study Chair — HIBA - cirugía pediátrica; Hernan Garcia Rivello, MD, Study Chair — HIBA - patología clínica; Marcelo Risk, PhD, Study Chair — IMTIB; Marcelo Rugiero, MD, Study Chair — HIBA - neurología; Julio Busaniche, MD, Study Chair — HIBA - clínica pediátrica; Rodolfo Pizarro, MD, Study Chair — HIBA - cardiología
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided
There is a plan to make individual participant data (IPD) available to other researchers by contacting the IP (María Lourdes Posadas Martínez, Soledad Kleppe, Marcelo Martín Serra) with a letter of intent on the protocol to be carried out. If you agree, the protocol will be presented to the ethics committee and work will be carried out in accordance with current regulations.

REFERENCES:
- [Background] Griggs RC, Batshaw M, Dunkle M, Gopal-Srivastava R, Kaye E, Krischer J, Nguyen T, Paulus K, Merkel PA; Rare Diseases Clinical Research Network. Clinical research for rare disease: opportunities, challenges, and solutions. Mol Genet Metab. 2009 Jan;96(1):20-6. doi: 10.1016/j.ymgme.2008.10.003. Epub 2008 Nov 13. PMID 19013090
- [Background] Stoller JK. The Challenge of Rare Diseases. Chest. 2018 Jun;153(6):1309-1314. doi: 10.1016/j.chest.2017.12.018. Epub 2018 Jan 8. PMID 29325986
- [Background] Gliklich RE, Dreyer NA, Leavy MB, editors. Registries for Evaluating Patient Outcomes: A User's Guide [Internet]. 3rd edition. Rockville (MD): Agency for Healthcare Research and Quality (US); 2014 Apr. Report No.: 13(14)-EHC111. Available from http://www.ncbi.nlm.nih.gov/books/NBK208616/ PMID 24945055